CLINICAL TRIAL: NCT04970693
Title: A Phase II Single-arm Study of Furmonertinib Combined With Radiotherapy for Non-small Cell Lung Cancer With Oligoprogression After First-line EGFR-TKI Therapy
Brief Title: A Study of Furmonertinib Combined With Radiotherapy for Non-small Cell Lung Cancer With Oligoprogression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1079
Record Dates: First submitted 2021-06-26; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Non-small Cell Lung Cancer; Oligoprogressive
Keywords: non-small cell lung cancer; oligoprogressive; Furmonertinib combined with radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furmonertinib 80mg combined with radiotherapy (Experimental): This group will enroll NSCLC patients who are oligoprogressive after first/second generation EGFR-TKI therapy. These patients will receive furmonertinib 80mg combined with radiotherapy as following therapy.
  Interventions: Drug: Furmonertinib
- Furmonertinib 160mg combined with radiotherapy (Experimental): This group will enroll NSCLC patients who are oligoprogressive after third generation EGFR-TKI therapy. These patients will receive furmonertinib 160mg combined with radiotherapy as following therapy.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — The different dose of furmonertinib will be given according to the generation of EGFR-TKI used as the first-line therapy. The doses and target volume of radiotherapy will be decided according to the oligoprogressive sites.
  Other Names: Radiotherapy

SUMMARY:
This Phase II randomized study is to explore the efficacy and safety of Furmonertinib combined with radiotherapy for non-small cell lung cancer with oligoprogression after first-line EGFR-TKI therapy.

DETAILED DESCRIPTION:
This Phase II randomized study is to explore the efficacy and safety of Furmonertinib combined with radiotherapy for non-small cell lung cancer with oligoprogression after first-line EGFR-TKI therapy.

The first group will enroll NSCLC patients with oligoprogression after using the first/second generation EGFR-TKI. The participants will receive Furmonertinib 80mg and local radiotherapy as the following therapy.

The other group will enroll NSCLC patients with oligoprogression after using the third generation EGFR-TKI. The participants will receive Furmonertinib 160mg and local radiotherapy as the following therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic NSCLC who are diagnosed by histology or cytology and are not suitable for surgery or radiotherapy;
* After receiving the first or second generation of EGFR-TKI treatment, the disease is oligoprogressive with 3-5 lesions (with imaging evidence), and the mutation is T790M+ (histological or hematological specimens, ARMS detection method);
* After receiving osimertinib treatment in the past, the disease is oligoprogressive with 3-5 lesions (with imaging evidence), and the patient refused chemotherapy;
* 18-80 years old;
* ECOG PS 0-2 scores;
* Organ and bone marrow functions were generally normal within 30 days before enrollment, including:AST, ALT ≤ 2.5 × ULN or ≤ 5 × ULN (with liver metastasis); total bilirubin ≤ 1.5 × ULN; neutrophils absolute value ≥ 1500 cells/mm3; Creatinine clearance ≥45 mL/min; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥90g/L.
* The baseline has measurable lesions defined by the RECIST 1.1 standard, and the progressive lesions should be treated with local radiotherapy; the definition of the lesion number includes:

  1. When there are lesions on both adrenal glands, it is considered to be 2 metastases;
  2. Two consecutive vertebral lesions and a paravertebral lesion within 6 cm can be considered as one metastasis, and the non-contiguous vertebral lesions should be counted separately;
  3. The adjacent lesions in the liver, lung, and mediastinum can be considered as a metastasis if one isocenter can be used for irradiation;
  4. Intracranial lesions are counted as 1 metastasis.
* The patient signed an informed consent form.

Exclusion Criteria:

* Severe or uncontrolled hypertension, diabetes, coronary artery stenosis, aortic dissection, aneurysm or acute bleeding disease;
* Any situation that increases the risk of QTc prolongation or arrhythmia;
* Left ventricular ejection fraction <50%;
* History of interstitial lung disease;
* FEV1%<30% or DLCO%<40%;
* Insertion of EGFR exon 20;
* The researcher believes that the patient is inappropriate to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2-year
  From the first day of treatment to the day of progression or the day of death.

SECONDARY OUTCOMES:
Overall survival | 2-year
  It was calculated from the first day of treatment to the day of death.
Failure pattern | 2-year
  Disease progression such as local recurrence or distant metastasis.
Safety evaluation | 2 year after therapy
  Adverse effects are graded according to the CTCAE 5.0 version, including multiple organs and tissues, such as gastrointestinal disease and symptom, cardiovascular disease, respiratory diseases and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Yu HA, Sima CS, Huang J, Solomon SB, Rimner A, Paik P, Pietanza MC, Azzoli CG, Rizvi NA, Krug LM, Miller VA, Kris MG, Riely GJ. Local therapy with continued EGFR tyrosine kinase inhibitor therapy as a treatment strategy in EGFR-mutant advanced lung cancers that have developed acquired resistance to EGFR tyrosine kinase inhibitors. J Thorac Oncol. 2013 Mar;8(3):346-51. doi: 10.1097/JTO.0b013e31827e1f83. PMID 23407558
- [Background] Schmid S, Klingbiel D, Aeppli S, Britschgi C, Gautschi O, Pless M, Rothschild S, Wannesson L, Janthur W, Foerbs D, Demmer I, Jochum W, Fruh M. Patterns of progression on osimertinib in EGFR T790M positive NSCLC: A Swiss cohort study. Lung Cancer. 2019 Apr;130:149-155. doi: 10.1016/j.lungcan.2019.02.020. Epub 2019 Feb 19. PMID 30885336
- [Background] Shah R, Lester JF. Tyrosine Kinase Inhibitors for the Treatment of EGFR Mutation-Positive Non-Small-Cell Lung Cancer: A Clash of the Generations. Clin Lung Cancer. 2020 May;21(3):e216-e228. doi: 10.1016/j.cllc.2019.12.003. Epub 2019 Dec 20. PMID 32014348
- [Background] Mu Y, Hao X, Xing P, Hu X, Wang Y, Li T, Zhang J, Xu Z, Li J. Acquired resistance to osimertinib in patients with non-small-cell lung cancer: mechanisms and clinical outcomes. J Cancer Res Clin Oncol. 2020 Sep;146(9):2427-2433. doi: 10.1007/s00432-020-03239-1. Epub 2020 May 8. PMID 32385709
- [Background] Eide IJZ, Helland A, Ekman S, Mellemgaard A, Hansen KH, Cicenas S, Koivunen J, Gronberg BH, Brustugun OT. Osimertinib in T790M-positive and -negative patients with EGFR-mutated advanced non-small cell lung cancer (the TREM-study). Lung Cancer. 2020 May;143:27-35. doi: 10.1016/j.lungcan.2020.03.009. Epub 2020 Mar 12. PMID 32200138
- [Background] Qiu B, Liang Y, Li Q, Liu G, Wang F, Chen Z, Liu M, Zhao M, Liu H. Local Therapy for Oligoprogressive Disease in Patients With Advanced Stage Non-small-cell Lung Cancer Harboring Epidermal Growth Factor Receptor Mutation. Clin Lung Cancer. 2017 Nov;18(6):e369-e373. doi: 10.1016/j.cllc.2017.04.002. Epub 2017 Apr 12. PMID 28465010
- [Background] Weickhardt AJ, Scheier B, Burke JM, Gan G, Lu X, Bunn PA Jr, Aisner DL, Gaspar LE, Kavanagh BD, Doebele RC, Camidge DR. Local ablative therapy of oligoprogressive disease prolongs disease control by tyrosine kinase inhibitors in oncogene-addicted non-small-cell lung cancer. J Thorac Oncol. 2012 Dec;7(12):1807-1814. doi: 10.1097/JTO.0b013e3182745948. PMID 23154552
- [Background] Shi Y, Zhang S, Hu X, Feng J, Ma Z, Zhou J, Yang N, Wu L, Liao W, Zhong D, Han X, Wang Z, Zhang X, Qin S, Ying K, Feng J, Fang J, Liu L, Jiang Y. Safety, Clinical Activity, and Pharmacokinetics of Alflutinib (AST2818) in Patients With Advanced NSCLC With EGFR T790M Mutation. J Thorac Oncol. 2020 Jun;15(6):1015-1026. doi: 10.1016/j.jtho.2020.01.010. Epub 2020 Jan 30. PMID 32007598
- [Background] Shi Y, Hu X, Zhang S, Lv D, Wu L, Yu Q, Zhang Y, Liu L, Wang X, Cheng Y, Ma Z, Niu H, Wang D, Feng J, Huang C, Liu C, Zhao H, Li J, Zhang X, Jiang Y, Gu C. Efficacy, safety, and genetic analysis of furmonertinib (AST2818) in patients with EGFR T790M mutated non-small-cell lung cancer: a phase 2b, multicentre, single-arm, open-label study. Lancet Respir Med. 2021 Aug;9(8):829-839. doi: 10.1016/S2213-2600(20)30455-0. Epub 2021 Mar 26. PMID 33780662